CLINICAL TRIAL: NCT05779527
Title: A Single Case Experimental Design Study of an Online Mindful-parenting Intervention for Parents of Children Living With a Visible Difference
Brief Title: Mindful Parenting - A Single Case Experimental Design Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiff University (Other)
Collaborators: University of Canterbury (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC.22.08.09.6601R2
Record Dates: First submitted 2022-12-20; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-01

CONDITIONS: Parenting; Alopecia; Skin Condition; Limb Difference; Neurofibromatoses; Craniofacial; Cleft Lip and Palate
MeSH Terms: conditions — Alopecia; Skin Diseases; Neurofibromatoses; Cleft Lip

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Mindful Parenting Programme (Experimental): Parents or carers will be invited to complete a six week online mindful parenting programme comprising online video, audio and written content plus four group support sessions via videoconferencing.
  Interventions: Behavioral: Mindful Parenting Programme

INTERVENTIONS:
Behavioral: Mindful Parenting Programme — Online Mindful Parenting Programme with group support sessions
  Other Names: Two Hearts

SUMMARY:
Some parents of children living with a visible difference can experience heightened stress due to the associated challenges of this. Parent's views of the child's visible difference and their responses to the child are important. Mindful parenting approaches have been found to reduce stress or distress for parents of children with disabilities, physical health problems and skin conditions.

This study will be completed with a small number of participants (around six to 12). Participants will be parents or carers of a child living with a visible difference aged four to 16 years, who are experiencing stress. Parents or carers will complete an online mindful parenting intervention (called Two Hearts) including video content, audio files and a workbook, over six weeks. Over the twelve-week study period participants will also provide the following information which will be compared over time:

* Complete four group support sessions during the intervention via videoconferencing
* Complete questionnaires at four timepoints
* Provide information about their use of the intervention materials and home practice weekly
* Answer two questions daily via text message about parenting stress levels We hope to learn about the initial effects of the mindful parenting programme for parents or carers of children living with a visible difference. We also hope to learn whether parents or carers find completing an online programme possible and practical. Finally, we hope to learn what parents' or carers' views are of the online programme and whether this type of intervention in online format would be helpful for other parents or carers.

DETAILED DESCRIPTION:
Aims

* To investigate the feasibility, acceptability, and initial effects of an online mindful parenting intervention for parents of children living with a visible difference.
* To investigate whether the intervention reduces parenting stress.
* To investigate whether completion of the intervention results in increased levels of mindful parenting.
* To investigate whether completion of the mindful parenting intervention has an impact upon child wellbeing.
* To investigate the feasibility of an online mindful parenting intervention for parents of children living with a visible difference, including adherence to the intervention, attrition, and participant perceptions of the acceptability of the intervention.

Hypotheses

* Completion of the intervention will result in changes in idiographic measures of parental stress. Namely, an improvement in the positive target and a reduction in the negative target. These improvements will be maintained on follow up.
* Completion of the intervention will result in reductions of parental stress on standardised assessment measures. These improvements will be maintained on follow up.
* Completion of the intervention will result in an improvement in child wellbeing on standardised assessment measures. These improvements will be maintained on follow up.
* Completion of the intervention will increase levels of mindful parenting as measured using a standardised assessment measure. These improvements will be maintained on follow up.
* Increased levels of mindful parenting will be associated with improved outcomes on idiographic and standardised assessment measures.

Methodology Design This study will adopt an A-B-A2 single case experimental design . Phase A will consist of a two-week baseline period. Phase B will be the six-week intervention. Phase A2 will be a four-week follow up period and an exit interview. The main outcome variable will be general parenting stress and parenting stress associated with the child's visible difference, measured idiographically via daily text messages. Secondary outcome variables will comprise standardised assessment measures of mindful parenting, parenting stress and parent reported child wellbeing. Feasibility of the online intervention will be assessed through recording of practical issues such as access to online content, participant adherence to the intervention (including home practice) and participant retention. Acceptability of the intervention will be assessed via participant evaluations of the workbook, online content, home practice and intervention overall through weekly feedback and the exit interview.

Participants The aim will be to recruit between six and 12 participants. Single case series methodology usually comprises only a small number of participants as each participant acts as their own control and provide large amounts of data.

Screening interview All participants will complete a screening interview to assess suitability for the intervention. During the screening interview the participants will be asked about 1. The nature of their child's visible difference, 2. Their access to a tablet or computer to complete the intervention, 3. Whether the parent is currently accessing any psychological therapy, 4. Parental mental health and stress (current and over the past year) including the use of medications, 5. Parental experience of mindfulness or meditation. Information obtained from the screening interview will be used to assess eligibility for the study, based on the above criteria.

Measures Demographic data Demographic information will be gathered at the beginning of the study. Parents will be asked to report their age, gender, ethnicity, education background; as well as their child's age, gender and nature of the visible difference (i.e. skin condition, mark, injury etc.) and part of the child's body affected.

Daily Idiographic measures of parenting stress Two unique targets identified by each participant around parenting stress will be measured daily on a scale of 1-100.

Standardised assessment measures Participants will be asked to complete standardised questionnaire measures at four timepoints: on baseline, immediately prior to beginning the intervention, immediately on completion and at follow up (four weeks after intervention completion).

Intervention engagement, home practice and retention Adherence and attrition will be recorded. Weekly feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice.

Intervention evaluation The acceptability of the intervention will be assessed through the following. An evaluation questionnaire will be used to assess parents' experiences of the Two Hearts Mindful Parenting intervention based on those developed by Bogels and Restifo for their Mindful Parenting programme. Parents will also complete an exit interview. Exit interviews will be audio recorded, or notes will be taken in line with participant preference. Where interviews are recorded these will be transcribed verbatim within six weeks of completion and then deleted.

Procedure Participants will first be interviewed via telephone to assess suitability. If the participant is suitable for the intervention, they will be directed to the online consent forms. If the participant choses to participate, then the researcher will support the parent to identify two target idiographic measures of parenting stress. A secure online text messaging service will be used to collect these measures from parents daily from baseline. Participants will be asked to complete standardised assessment measures through the online platform Qualtrics at four timepoints (baseline, immediately prior to starting the intervention, immediately on completion of the intervention and at four week follow up). Participants will be asked to provide weekly feedback regarding their engagement with the intervention materials and home practice. Participants will be able to begin the online intervention when enough participants have been recruited and at least two weeks after they complete their baseline measures. On completion of the follow up period participants will be asked to complete an exit interview.

Recruitment strategy Charitable foundations such as Changing Faces, Cleft Lip and Palate Association (CLAPA), the Children's Burns Trust (CBT), Headlines Craniofacial Support, and Ichthyosis Support Group, based in the UK, will be invited to share our recruitment advert and a link to our study information sheet on their social media pages and websites. Snowball sampling will be enabled to allow wide distribution.

Intervention The Two Hearts mindful parenting is an online programme based on the Mindful Parenting programme developed by Bogels & Restifo and was developed by an expert panel (L-M. Emerson, S. Bögels, J. Paynter). The intervention has been piloted with parents from a community population. In this pilot study the intervention was found to be acceptable to parents. Intervention retention was 100%, however adherence to home practice was variable. Reductions in parenting stress and increased levels of mindfulness were reported for half of the participants. The Mindful Parenting intervention will be free for participants. Parents only will complete the intervention.

The Two Hearts programme comprises four self-directed online modules, which involve video and audio recorded content supported by a parent workbook (Introduction, Mindful Awareness in Parenting, Mindful Parenting in Action, Compassion in Parenting). The introductory module will consist of a brief PDF document alongside an audio file to support home practice. All three other modules consist of a series of two to four short videos to be accessed via an appropriate online platform, reading from the Parent Workbook and audio files to support mindfulness practices. Mindfulness practices include three-minute breathing space and mindful movement.

The intervention period will begin when enough participants have been recruited and around two-weeks after participants complete baseline measures. Intervention content is to be hosted on an online platform and parents will be able to access one module at a time over the six-week intervention period. Participants will be encouraged to engage in regular mindfulness home practice.

Participants will be supported to engage with the intervention via text message reminders twice a week during the six-week intervention period and once per week during the four-week follow up period. Four group support sessions (videoconferencing) will be scheduled at the start of the programme (introduction) after week two, week four and week six. These sessions will be organised with participants in small groups (or individually if necessary). Participants will be sent a link to the group support sessions via email. Sessions will be conducted via videoconferencing. No data will be collected during these sessions other than attendance data, and they will not be recorded. At the beginning of group support sessions issues of confidentiality (and it's limits) and group conduct will be discussed. Support sessions are intended to help participants overcome any barriers to engaging with the intervention materials or completing home practice. Attendance data will be linked with anonymised participant numbers on a secure database.

Data Analysis

Idiographic data:

Idiographic data will be organised in excel and observed in a graph and analysed visually to identify trends, variability and data patterns.

Idiographic data will be analysed with Tau-U via an online calculator. Tau-U examines data non-overlap between study phases (baseline, intervention, follow-up). Baseline scores will initially be analysed for trend and any significant trend will be corrected for. Weighted averages will be calculated.

Secondary outcome data:

Differences between phases (baseline, intervention, and follow up) on secondary outcome measures will be examined using Jacobson's reliable change index. The distribution of scores on these measures will be gathered from existing literature to generate reliable change criteria. Analyses will be completed employing the Leeds Reliable Change Indicator .

Evaluation data:

Quantitative intervention engagement data, evaluation form data and exit interview data will be tabulated. Descriptive analyses and frequencies will be reported. Thematic analysis will be used to identify themes from qualitative exit interview data.

ELIGIBILITY:
Inclusion Criteria:

* Parents aged over 16 years, of children aged between four (4)-16 years living with a visible difference
* All types and aetiologies of child visible differences including any scarring, condition, disability, or mark that affects a person's appearance, with confirmation via self-report
* Parent experiencing self-reported stress associated with the child's visible difference
* Able to communicate in verbal and written English
* Access to a computer/tablet with an active internet connection

Exclusion Criteria:

* Parent currently accessing psychological therapy for their own wellbeing, including parenting programmes
* Parent experiencing active thoughts of suicide or self-injury
* Parent experienced a psychotic episode or engaged in deliberate self-injury over the past year
* Parent commenced medications for mood in the last two months
* Parent previously accessed a mindful parenting intervention
* Child currently in an acute phase following a physical injury
* Only one parent or carer per household can take part

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-03-28 (Estimated); Study Completion 2023-04-14 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress (unique to each participant) | Day 1
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 2
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 3
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 4
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 5
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 6
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 7
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 8
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 9
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 10
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 11
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 12
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 13
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 14
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 15
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 16
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 17
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 18
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 19
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 20
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 21
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 22
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 23
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 24
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 25
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 26
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 27
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 28
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 29
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 30
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 31
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 32
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 33
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 34
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 35
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 36
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 37
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 38
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 39
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 40
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 41
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 42
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 43
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 44
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 45
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 46
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 47
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 48
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 49
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 50
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 51
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 52
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 53
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 54
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 55
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 56
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 57
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 58
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 59
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 60
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 61
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 62
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 63
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 64
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 65
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 66
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 67
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 68
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 69
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 70
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 71
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 72
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 73
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 74
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 75
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 76
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 77
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 78
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 79
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 80
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 81
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 82
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 83
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.
Parenting Stress (unique to each participant) | Day 84
  Parents will identify two targets for desired change around parenting stress related to the child's visible difference. It is intended that participants will identify one target area for improvement (positive target) and one for reduction (negative target). Questions will be rated on a scale of 0 (not at all) to 100 (extremely). Idiographic measures will be completed via text message. Text messages will be sent via a secure online provider (PageOne's Janet txt). Example targets include: be more present in interactions with my child and be grumpy or respond abruptly with my child less.

SECONDARY OUTCOMES:
Parenting Stress Index 4th Edition Short Form | Baseline
  Measure of Parenting Stress with total stress reported on a scale of 36-180 and higher scores being indicative of higher levels of stress.
Parenting Stress Index 4th Edition Short Form | Pre-intervention (week 2)
  Measure of Parenting Stress with total stress reported on a scale of 36-180 and higher scores being indicative of higher levels of stress.
Parenting Stress Index 4th Edition Short Form | Post-intervention (week 8)
  Measure of Parenting Stress with total stress reported on a scale of 36-180 and higher scores being indicative of higher levels of stress.
Parenting Stress Index 4th Edition Short Form | Follow up (week 12)
  Measure of Parenting Stress with total stress reported on a scale of 36-180 and higher scores being indicative of higher levels of stress.
Interpersonal Mindfulness in Parenting scale | Baseline
  Measure of Mindful Parenting measured on a scale of 31-155 for total mindfulness with higher scores indicative of higher levels of mindful parenting.
Interpersonal Mindfulness in Parenting scale | Pre-intervention (week 2)
  Measure of Mindful Parenting measured on a scale of 31-155 for total mindfulness with higher scores indicative of higher levels of mindful parenting.
Interpersonal Mindfulness in Parenting scale | Post-intervention (week 8)
  Measure of Mindful Parenting measured on a scale of 31-155 for total mindfulness with higher scores indicative of higher levels of mindful parenting.
Interpersonal Mindfulness in Parenting scale | Follow up (week 12)
  Measure of Mindful Parenting measured on a scale of 31-155 for total mindfulness with higher scores indicative of higher levels of mindful parenting.
Strengths and Difficulties questionnaire (SDQ) | Baseline
  Parent reported child wellbeing measure with scores ranging from 0-40 with higher scores being indicative of higher levels of difficulty on all subscales other than the prosocial subscale.
Strengths and Difficulties questionnaire (SDQ) | Pre-intervention (week 2)
  Parent reported child wellbeing measure with scores ranging from 0-40 with higher scores being indicative of higher levels of difficulty on all subscales other than the prosocial subscale.
Strengths and Difficulties questionnaire (SDQ) | Post-intervention (week 8)
  Parent reported child wellbeing measure with scores ranging from 0-40 with higher scores being indicative of higher levels of difficulty on all subscales other than the prosocial subscale.
Strengths and Difficulties questionnaire (SDQ) | Follow up (week 12)
  Parent reported child wellbeing measure with scores ranging from 0-40 with higher scores being indicative of higher levels of difficulty on all subscales other than the prosocial subscale.

OTHER OUTCOMES:
Participant evaluation of the Mindful Parenting Programme | Follow up (week 12)
  An evaluation questionnaire will be used to assess parents' experiences of the Two Hearts Mindful Parenting intervention based on those developed by previous authors. Questions include: "Do you feel you've got something of lasting value of importance because of taking the training?", adherence to home practice "On average, how many times a week did you practice the meditation exercises during the course?", and perceived importance/ value of specific elements of the intervention "body scan".
Exit interview to gather feedback on participant experience of participation in the study | Follow up (week 12)
  Questions will include: "What was your experience of the video content of the intervention?", "What was your experience of the support sessions?", "Are there any practices in you plan to take forwards beyond the end of the study?", "Have you noticed any changes in their self-compassion?", and "What changes, if any, have you noticed in the way you interact with your child?".
Levels of participant engagement with intervention materials and home practice exercises | Week 3
  Adherence and attrition will be recorded. Feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice. Participants will provide this information via text message giving the number of minutes spent on each reading intervention materials and engaging with home practice.
Levels of participant engagement with intervention materials and home practice exercises | Week 4
  Adherence and attrition will be recorded. Feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice. Participants will provide this information via text message giving the number of minutes spent on each reading intervention materials and engaging with home practice.
Levels of participant engagement with intervention materials and home practice exercises | Week 5
  Adherence and attrition will be recorded. Feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice. Participants will provide this information via text message giving the number of minutes spent on each reading intervention materials and engaging with home practice.
Levels of participant engagement with intervention materials and home practice exercises | Week 6
  Adherence and attrition will be recorded. Feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice. Participants will provide this information via text message giving the number of minutes spent on each reading intervention materials and engaging with home practice.
Levels of participant engagement with intervention materials and home practice exercises | Week 7
  Adherence and attrition will be recorded. Feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice. Participants will provide this information via text message giving the number of minutes spent on each reading intervention materials and engaging with home practice.
Levels of participant engagement with intervention materials and home practice exercises | Week 8
  Adherence and attrition will be recorded. Feedback will be collected from participants regarding levels of engagement with the intervention and mindfulness home practice. Participants will provide this information via text message giving the number of minutes spent on each reading intervention materials and engaging with home practice.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Thompson, Principal Investigator — Cardiff University
Locations (1):
- Cardiff University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abidin, R. (2012). Parenting Stress Index-Fourth Edition (PSI-4). Lutz, FL: Psychological Assessment Resources.
- [Background] Bögels, S., & Restifo, K. (2013). Mindful parenting: A guide for mental health practitioners. Springer Science & Business Media.
- [Background] Dempsey L, Dowling M, Larkin P, Murphy K. Sensitive Interviewing in Qualitative Research. Res Nurs Health. 2016 Dec;39(6):480-490. doi: 10.1002/nur.21743. Epub 2016 Jul 19. PMID 27434172
- [Background] Emerson, L. M., Aktar, E., de Bruin, E., Potharst, E., & Bögels, S. (2019). Mindful Parenting in Secondary Child Mental Health: Key Parenting Predictors of Treatment Effects. Mindfulness, 1-11.
- [Background] Heapy C, Norman P, Emerson LM, Murphy R, Bogels S, Thompson AR. Mindful parenting intervention for parents of children with skin conditions: a single group experimental cases series. Behav Cogn Psychother. 2022 Sep;50(5):462-480. doi: 10.1017/S1352465822000170. Epub 2022 Apr 25. PMID 35466907
- [Background] Jacobson NS, Truax P. Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol. 1991 Feb;59(1):12-9. doi: 10.1037//0022-006x.59.1.12. PMID 2002127
- [Background] Kabat-Zinn, J. (2013). Full Catastrophe Living, Revised Edition: How to Cope with Stress, Pain and Illness Using Mindfulness Meditation: Hachette uK.
- [Background] Morley, S., & Dowzer, C. (2014). The Leeds Reliable Change Indicator. University of Leeds.
- [Background] Parker RI, Vannest KJ, Davis JL, Sauber SB. Combining nonoverlap and trend for single-case research: Tau-U. Behav Ther. 2011 Jun;42(2):284-99. doi: 10.1016/j.beth.2010.08.006. Epub 2011 Feb 3. PMID 21496513
- [Background] Sherwood, A. (2020). Mindful Parenting Brief Online Intervention: Exploring Program Feasibility and Initial Effects. Griffith University Gold Coast,
- [Background] Vannest, K. J., Parker, R. I., Gonen, O., & Adiguzel, T. (2016). Single Case Research: Web Based Calculators for Scr Analysis. Retrieved from http://www.singlecaseresearch.org/